CLINICAL TRIAL: NCT04569058
Title: Transcranial Photobiomodulation Therapy for the Treatment of Autistic Traits in Children and Adolescents With Attention Deficit Hyperactivity Disorder
Brief Title: Transcranial Photobiomodulation Therapy for the Treatment of Autistic Traits in Children and Adolescents With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Tolga A Ceranoglu, Associate Psychiatrist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-P-002352
Record Dates: First submitted 2020-09-18; First posted 2020-09-29 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: Autism; Attention Deficit Hyperactivity Disorder
Keywords: Autistic Traits; ADHD; Attention; Autism; photobiomodulation; transcranial light therapy
MeSH Terms: conditions — Autistic Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Transcranial Photobiomodulation (Experimental): Transcranial Photobiomodulation--a noninvasive intervention in which near-infrared light (850 nanometer) is applied to forebrain.
  Interventions: Device: Transcranial Photobiomodulation

INTERVENTIONS:
Device: Transcranial Photobiomodulation — Transcranial Photobiomodulation--a noninvasive intervention in which near-infrared light (850 nanometer) is applied to forebrain.
  Other Names: Niraxx G1 Headband

SUMMARY:
An open label trial to assess the safety and efficacy of transcranial photobiomodulation (tPBM) in improving autistic traits in ADHD youth.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder characterized by variable presentation of difficulties with socialization, reciprocal communication, and restrictive/repetitive behaviors. An increasingly higher prevalence of ASD is documented in each successive epidemiological survey and the disorder is now estimated to affect up to 2% of youth in the general population. This rise in prevalence is in part attributed to improved recognition of autism in intellectually capable populations.

There exists no established pharmacological treatment for the core features of ASD.

Current practice consists of well-established evidence-based pharmacotherapies that are available for the management of comorbid psychiatric disorders, in order to improve quality of life and reduce symptom severity in ASD. Clinical trials of available treatment options reveal that compared to general population, individuals with ASD may be more susceptible to adverse effects of medications which could be dose-related, and may have lower adherence to treatment. New treatments for core deficits in ASD are needed; an intervention requiring no medication may offer better compliance and tolerability.

Attention Deficit/Hyperactivity Disorder (ADHD) is the most common psychiatric disorder recognized in youth and adults with ASD, and greatly adds to their morbidity and dysfunction, particularly in those with intact intellectual capacity. The prevalence of ADHD in the general population of school-age children is approximately 3% to 5%, although some reports show even higher incidence. Nearly two-thirds of referred populations of youth (ranging from 59-83%) and adults (ranging from 37-68%) with ASD suffer from ADHD.

Both ADHD and ASD have strong shared heritable components according to the evidence from twin and family studies. Up to 15% of youth with ADHD suffer from ASD and experience greater morbidity and dysfunction. This confounding effect of ASD seems to be symptom dependent and not contingent upon reaching full diagnostic threshold. In fact, up to a third of ADHD youth without ASD diagnosis still struggle with persistent symptoms of ASD (henceforth termed autistic traits [ATs]) and associated compromised outcomes. Presence of ATs is associated with a more complicated course of ADHD, characterized as increased comorbid psychopathology, more impaired interpersonal, school, family, and cognitive functioning. Anti-ADHD medications effectively mitigate core symptoms of ADHD, but offer no improvement in the ATs. Youth with ADHD continue to suffer from the impairments associated with ATs that prognosticate a compromised course in multiple domains of functioning despite effective treatment of ADHD. Treating comorbid ATs in patients with ADHD could prevent functional deterioration, and improve long term outcomes. As yet, there exists no known treatment for the core features of ASD or ATs.

A novel treatment approach for social and cognitive deficits is based on transcranial application of Light Emitting Diode (LED), an invisible, non-ionizing electromagnetic wave. Referred to as Transcranial Photobiomodulation, tPBM consists of exposing bilaterally the frontal brain to a non-ionizing electromagnetic wave. The transcranial photobiomodulation (tPBM) is invisible, penetrates the skin and skull into brain tissue, is non-invasive, and minimally dissipated as thermal energy. The benefits of tPBM are wavelength specific. A mitochondrial enzyme, the cytochrome c oxidase, is the primary chromophore for the tPBM at wavelengths of 830-850 nanometers. What follows is, increased adenosine triphosphate (ATP) production, through the respiratory chain. Ultimately, the increased ATP leads to increased energy metabolism for the cell, and it is hypothesized that a signaling cascade is also activated promoting cellular plasticity and cytoprotection.

Unique properties of the tPBM have led to novel therapeutic applications in neurology, for treatment following acute ischemic stroke subjects, and in dermatology for treatment of alopecia. In psychiatric care, tPBM has been shown to be safe, effective and well tolerated compared the sham treatment in patients with Major Depressive Disorder (MDD).

These properties of the tPBM have led to novel therapeutic applications in neurology. In acute ischemic stroke subjects, acute treatment with the tPBM led to significantly better outcome as compared to sham. These results were confirmed in a different cohort of stroke patients with mild to moderate severity of illness. Both studies on stroke subjects showed no significant difference in rate of adverse events, as well as serious adverse events, between the tPBM and sham treated subjects. The tPBM has also been used as a treatment of alopecia and in animal models for methanol-induced retinal toxicity. The tPBM is already widely used for non-invasive assessment of brain function (replacing functional magnetic resonance imaging in studies of infants and young adults, under the name of Near Infrared Spectroscopy) underscoring the relatively low risk of tPBM.

Proposed treatment with tPBM has been previously studied in patients with Major Depressive Disorder (MDD). MDD has been associated with deficits in brain bioenergetic metabolism. In an experimental model of depression, the mitochondrial respiratory chain (the cellular site for energy production) was found to be inhibited by chronic stress. Depressed subjects have also significantly lower production of ATP (an energy vector) in their muscle tissue and greater incidence of deletions in their mitochondrial DNA. Data from magnetic resonance spectroscopy in subjects with MDD showed that response to the augmentation of a selective serotonin reuptake inhibitor (SSRI) with triiodothyronine (a thyroid hormone) is associated with restoration of the levels of ATP in the brain. A preliminary open study in 10 depressed subjects has shown that the tPBM was safe, effective and well tolerated.

More recently, a proof of concept study was conducted with tPBM, in an open label, prospective design with 10 patients with a diagnosis of ASD between ages 18 and 55. Five patients met the rigorous responder criteria, and a statistically significant improvement was observed in all clinician and patient rated measures at midpoint and endpoint. Efficacy measures revealed that tPBM substantially improved ATs in 7 patients (70%), and was well tolerated with no treatment-limiting side-effects or serious adverse events. Adherence rate among participants was 98%.

These findings suggest that tPBM may be a promising treatment for core social deficits associated with ASD and is a safe, feasible treatment approach. The major risk of tPBM when using a laser as the light source is associated with accidental retinal exposure, when beams are projected through the lens, with increased risk of macular degeneration. LED light does not share the same risk level as laser light sources. Based on these promising results, this novel treatment approach is safe, well-tolerated and associated with statistically and clinically significant improvements in symptoms of ASD.

The researchers hypothesize that tPBM will be safe and effective in the treatment of ATs in youth with ADHD, and will improve social functioning, which stimulants do not address.

Aforementioned proof-of-concept study was blessed with a fast pace of recruitment, with 10 participants over a period of 18 months, despite its demanding nature for our patients. Even faster and more efficient recruitment along with a less demanding schedule for our patients is possible. Telemedicine substitutes for face-to-face office visits through a remote, two-way video-conference through secure Internet access. Telemedicine use in the clinical setting has successfully provided specialist advice with favorable patient outcomes, satisfaction, and costs. Clinical trials are the gold standard for evaluating new therapeutic opportunities in medicine, efforts aimed at improving their efficiency are needed to facilitate patient participation in a manner that reduces dropout, and Telemedicine may offer such opportunity.

The researchers propose an open label trial to assess the safety and efficacy of tPBM in improving ATs in ADHD youth with comorbid ATs. Eligible participants will be youth with adequately treated ADHD who present with comorbid ATs of at least moderate severity. Participants will receive tPBM daily for 8 weeks. Participants who meet eligibility criteria will be mailed the tPBM device. They will be able to administer the treatment in the comfort of home, at scheduled intervals. Accurate application of tPBM, its safety, and efficacy will be assessed during regular scheduled meetings with study clinician. These meetings will all be conducted via telemedicine with HIPAA compliant communication technology. Safety of and treatment response to tPBM will be monitored by parent- and clinician-rated measures during regularly scheduled visits. The study will address the question whether tPBM is effective for the treatment of ATs in youth with ADHD, and whether it is acceptable among our patients.

Certain aspects of tPBM render it a feasible intervention. It can be delivered at home. It does not require ingestion of any substances. It is possible that the exposure to tPBM might be more acceptable than use of medications among some minority groups. This intervention does not require providers with specific cultural expertise or second language proficiency.

The tPBM treatment can be completed in the comfort of participants' homes, while monitoring their safety and response during scheduled medicine visits. The advantage of the tPBM treatment approach compared to pharmacotherapy is that adherence can be easily monitored. This study will answer whether tPBM has an effect on ASD symptoms in ADHD and whether it is acceptable among our patients, for whom frequent visits otherwise would be prohibitive or render it inaccessible. As such, the researchers propose the inclusion of a telemedicine visits in this study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants between 9 and 17 years of age (inclusive)
* Participant fulfills Diagnostic and Statistical Manual of Mental Disorders-5 diagnostic criteria for Attention Deficit Hyperactivity Disorder as established by the clinical diagnostic interview.
* Participants with at least moderate severity of Autism Spectrum Disorder symptoms as demonstrated by Social Responsiveness Scale raw score ≥ 75 or Clinician Global Impression-Autistic Traits severity score ≥ 4
* Participants must understand the nature of the study. Participants must sign an Institutional Review Board-approved informed consent form before initiation of any study procedures.
* Participants are willing and able to cooperate with all tests, examinations and demonstrate ability to appropriately administer the study treatment required by the protocol.
* Participants must have access to a computer with camera and broadband internet connection

Exclusion Criteria:

* Impaired intellectual capacity (clinically determined)
* Serious chronic medical or psychiatric condition that, in the investigator's opinion, puts the subject at risk
* The subject has a significant skin condition at the procedure sites (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo)
* The subject has an implant of any kind in the head (e.g. stent, clipped aneurysm, embolised AVM, implantable shunt - Hakim valve)
* Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment including: Visudine (verteporfin) - for age related macular degeneration; Aminolevulinic Acid- for actinic keratoses; Photofrin (porfimer sodium) - for esophageal cancer, non-small cell lung cancer; Levulan Kerastick (aminolevulinic acid HCl) - for actinic keratosis; 5-aminolevulinic acid; and (ALA)- for non-melanoma skin cancer
* Current treatment with a psychotropic medication on a dose that has not been stable for at least 4 weeks prior to initiating study treatment.
* Pregnant or nursing females
* Investigator and his/her immediate family

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: T. Atilla Ceranoglu, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blumberg SJ, Bramlett MD, Kogan MD, Schieve LA, Jones JR, Lu MC. Changes in prevalence of parent-reported autism spectrum disorder in school-aged U.S. children: 2007 to 2011-2012. Natl Health Stat Report. 2013 Mar 20;(65):1-11, 1 p following 11. PMID 24988818
- [Background] Joshi G, Petty C, Wozniak J, Henin A, Fried R, Galdo M, Kotarski M, Walls S, Biederman J. The heavy burden of psychiatric comorbidity in youth with autism spectrum disorders: a large comparative study of a psychiatrically referred population. J Autism Dev Disord. 2010 Nov;40(11):1361-70. doi: 10.1007/s10803-010-0996-9. PMID 20309621
- [Background] Campbell M, Fish B, David R, Shapiro T, Collins P, Koh C. Response to triiodothyronine and dextroamphetamine: a study of preschool schizophrenic children. J Autism Child Schizophr. 1972 Oct-Dec;2(4):343-58. doi: 10.1007/BF01538168. No abstract available. PMID 4581614
- [Background] Stigler KA, Desmond LA, Posey DJ, Wiegand RE, McDougle CJ. A naturalistic retrospective analysis of psychostimulants in pervasive developmental disorders. J Child Adolesc Psychopharmacol. 2004 Spring;14(1):49-56. doi: 10.1089/104454604773840481. PMID 15142391
- [Background] Handen BL, Johnson CR, Lubetsky M. Efficacy of methylphenidate among children with autism and symptoms of attention-deficit hyperactivity disorder. J Autism Dev Disord. 2000 Jun;30(3):245-55. doi: 10.1023/a:1005548619694. PMID 11055460
- [Background] Joshi G, Biederman J, Petty C, Goldin RL, Furtak SL, Wozniak J. Examining the comorbidity of bipolar disorder and autism spectrum disorders: a large controlled analysis of phenotypic and familial correlates in a referred population of youth with bipolar I disorder with and without autism spectrum disorders. J Clin Psychiatry. 2013 Jun;74(6):578-86. doi: 10.4088/JCP.12m07392. PMID 23842009
- [Background] Stahlberg O, Soderstrom H, Rastam M, Gillberg C. Bipolar disorder, schizophrenia, and other psychotic disorders in adults with childhood onset AD/HD and/or autism spectrum disorders. J Neural Transm (Vienna). 2004 Jul;111(7):891-902. doi: 10.1007/s00702-004-0115-1. PMID 15206005
- [Background] Polanczyk G, de Lima MS, Horta BL, Biederman J, Rohde LA. The worldwide prevalence of ADHD: a systematic review and metaregression analysis. Am J Psychiatry. 2007 Jun;164(6):942-8. doi: 10.1176/ajp.2007.164.6.942. PMID 17541055
- [Background] de Bruin EI, Ferdinand RF, Meester S, de Nijs PF, Verheij F. High rates of psychiatric co-morbidity in PDD-NOS. J Autism Dev Disord. 2007 May;37(5):877-86. doi: 10.1007/s10803-006-0215-x. PMID 17031447
- [Background] Leyfer OT, Folstein SE, Bacalman S, Davis NO, Dinh E, Morgan J, Tager-Flusberg H, Lainhart JE. Comorbid psychiatric disorders in children with autism: interview development and rates of disorders. J Autism Dev Disord. 2006 Oct;36(7):849-61. doi: 10.1007/s10803-006-0123-0. PMID 16845581
- [Background] Mattila ML, Hurtig T, Haapsamo H, Jussila K, Kuusikko-Gauffin S, Kielinen M, Linna SL, Ebeling H, Bloigu R, Joskitt L, Pauls DL, Moilanen I. Comorbid psychiatric disorders associated with Asperger syndrome/high-functioning autism: a community- and clinic-based study. J Autism Dev Disord. 2010 Sep;40(9):1080-93. doi: 10.1007/s10803-010-0958-2. PMID 20177765
- [Background] Sinzig J, Walter D, Doepfner M. Attention deficit/hyperactivity disorder in children and adolescents with autism spectrum disorder: symptom or syndrome? J Atten Disord. 2009 Sep;13(2):117-26. doi: 10.1177/1087054708326261. Epub 2009 Apr 20. PMID 19380514
- [Background] Autism and Developmental Disabilities Monitoring Network Surveillance Year 2002 Principal Investigators; Centers for Disease Control and Prevention. Prevalence of autism spectrum disorders--autism and developmental disabilities monitoring network, 14 sites, United States, 2002. MMWR Surveill Summ. 2007 Feb 9;56(1):12-28. PMID 17287715
- [Background] Christensen DL, Maenner MJ, Bilder D, Constantino JN, Daniels J, Durkin MS, Fitzgerald RT, Kurzius-Spencer M, Pettygrove SD, Robinson C, Shenouda J, White T, Zahorodny W, Pazol K, Dietz P. Prevalence and Characteristics of Autism Spectrum Disorder Among Children Aged 4 Years - Early Autism and Developmental Disabilities Monitoring Network, Seven Sites, United States, 2010, 2012, and 2014. MMWR Surveill Summ. 2019 Apr 12;68(2):1-19. doi: 10.15585/mmwr.ss6802a1. PMID 30973853
- [Background] Fombonne E. Epidemiological surveys of autism and other pervasive developmental disorders: an update. J Autism Dev Disord. 2003 Aug;33(4):365-82. doi: 10.1023/a:1025054610557. PMID 12959416
- [Background] Kogan MD, Blumberg SJ, Schieve LA, Boyle CA, Perrin JM, Ghandour RM, Singh GK, Strickland BB, Trevathan E, van Dyck PC. Prevalence of parent-reported diagnosis of autism spectrum disorder among children in the US, 2007. Pediatrics. 2009 Nov;124(5):1395-403. doi: 10.1542/peds.2009-1522. Epub 2009 Oct 5. PMID 19805460
- [Background] Ronald A, Happe F, Bolton P, Butcher LM, Price TS, Wheelwright S, Baron-Cohen S, Plomin R. Genetic heterogeneity between the three components of the autism spectrum: a twin study. J Am Acad Child Adolesc Psychiatry. 2006 Jun;45(6):691-699. doi: 10.1097/01.chi.0000215325.13058.9d. PMID 16721319
- [Background] Joshi G, Faraone SV, Wozniak J, Tarko L, Fried R, Galdo M, Furtak SL, Biederman J. Symptom Profile of ADHD in Youth With High-Functioning Autism Spectrum Disorder: A Comparative Study in Psychiatrically Referred Populations. J Atten Disord. 2017 Aug;21(10):846-855. doi: 10.1177/1087054714543368. Epub 2014 Aug 1. PMID 25085653
- [Background] Mochizuki-Oda N, Kataoka Y, Cui Y, Yamada H, Heya M, Awazu K. Effects of near-infra-red laser irradiation on adenosine triphosphate and adenosine diphosphate contents of rat brain tissue. Neurosci Lett. 2002 May 3;323(3):207-10. doi: 10.1016/s0304-3940(02)00159-3. PMID 11959421
- [Background] Lampl Y, Zivin JA, Fisher M, Lew R, Welin L, Dahlof B, Borenstein P, Andersson B, Perez J, Caparo C, Ilic S, Oron U. Infrared laser therapy for ischemic stroke: a new treatment strategy: results of the NeuroThera Effectiveness and Safety Trial-1 (NEST-1). Stroke. 2007 Jun;38(6):1843-9. doi: 10.1161/STROKEAHA.106.478230. Epub 2007 Apr 26. PMID 17463313
- [Background] Cassano P, Cusin C, Mischoulon D, Hamblin MR, De Taboada L, Pisoni A, Chang T, Yeung A, Ionescu DF, Petrie SR, Nierenberg AA, Fava M, Iosifescu DV. Near-Infrared Transcranial Radiation for Major Depressive Disorder: Proof of Concept Study. Psychiatry J. 2015;2015:352979. doi: 10.1155/2015/352979. Epub 2015 Aug 19. PMID 26356811
- [Background] Cassano P, Petrie SR, Hamblin MR, Henderson TA, Iosifescu DV. Review of transcranial photobiomodulation for major depressive disorder: targeting brain metabolism, inflammation, oxidative stress, and neurogenesis. Neurophotonics. 2016 Jul;3(3):031404. doi: 10.1117/1.NPh.3.3.031404. Epub 2016 Mar 4. PMID 26989758
- [Background] Schiffer F, Johnston AL, Ravichandran C, Polcari A, Teicher MH, Webb RH, Hamblin MR. Psychological benefits 2 and 4 weeks after a single treatment with near infrared light to the forehead: a pilot study of 10 patients with major depression and anxiety. Behav Brain Funct. 2009 Dec 8;5:46. doi: 10.1186/1744-9081-5-46. PMID 19995444

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants ages 9-17: Participants ages 9-17 enrolled to receive tPBM treatment.
Period: Overall Study
Arm/Group | Participants ages 9-17
Started | 38
Completed | 31
Not Completed | 7

BASELINE CHARACTERISTICS:
Population: Seven participants were excluded from the analysis.
Arm/Group | Participants Ages 9-17
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants] — Population: Seven participants were excluded from the analysis
  Participants
    <=18 years | 31
    Between 18 and 65 years | 0
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Seven participants were excluded from the analysis
  Participants
    Female | 7
    Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Seven participants were excluded from the analysis
  Participants
    Hispanic or Latino | 4
    Not Hispanic or Latino | 27
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Seven participants were excluded from the analysis
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 24
    More than one race | 1
    Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Symptom Checklist (ADHD-SCL)
Description: The ADHD-SCL is a clinician-rated scale used to determine the number and severity of ADHD symptoms that a patient may be experiencing. It consists of 18 items that rated on a scale from 0 (no symptoms) to 3 (severe symptoms). The item scores are combined into a total score which ranges from 0 to 54, where a higher score indicates a worse outcome. The outcome reported reflects the change from baseline in ADHD-SCL scores and negative scores represent improvement (i.e., decrease in severity from baseline).
Time Frame: Baseline to week 8
Population: Participants who were exposed to study treatment for at least two weeks.
Measure: Mean (Standard Deviation); unit: change in scale score
Groups:
- tPBM treatment: Participants who received tPBM treatment
Arm/Group | tPBM treatment
Number analyzed (Participants) | 31
change in scale score | -8.5 (8.8)

2. Primary Outcome: Change From Baseline in Social Responsiveness Scale-2 (SRS-2)
Description: The SRS-2 is a parent-rated scale used to identify the presence and severity of social impairment within the autism spectrum and differentiate it from that which occurs in other disorders. It consists of 65 items that rated on a scale from 1 (not true) to 4 (almost always true). Items are combined into a total score which ranges from 0 to 195, where a higher score indicates a worse outcome. The outcome reported reflects the change from baseline in SRS Total raw scores and negative scores represent improvement (i.e., decrease in severity from baseline).
Time Frame: Baseline to week 8
Population: Participants who were exposed to study treatment for at least two weeks.
Measure: Mean (Standard Deviation); unit: change in scale score
Arm/Group | tPBM treatment
Number analyzed (Participants) | 31
change in scale score | -25.5 (26.4)

3. Secondary Outcome: Level of Discomfort at Study Endpoint Measured by the Transcranial Photobiomodulation Self-Report Questionnaire (TSRQ)
Description: The TSRQ is a patient-rated scale used to assess the safety of transcranial photobiomodulation for treatment of autistic traits in youth with ADHD. It consists of 5 items, with the first item assessing patient discomfort during the transcranial photobiomodulation on a scale of 0 (no discomfort) to 5 (extreme discomfort). The outcome reported reflects the number of patients who experienced each discomfort level at the last study visit.
Time Frame: Week 8 (study endpoint)
Population: Participants who were exposed to study treatment for at least two weeks.
Measure: Number; unit: participants
Arm/Group | tPBM treatment
Number analyzed (Participants) | 31
participants
  No discomfort at study end point | 27
  Mild discomfort at study end point | 4
  Moderate discomfort at study end point | 0
  Severe discomfort at study end point | 0
  Extreme discomfort at study end point | 0

ADVERSE EVENTS:
Time Frame: Adverse events in all participants who started treatment (baseline through week 10 follow-up visit)
Arm/Group | Participants ages 9-17
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 26/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants ages 9-17 (N=31)
Local/treatment site reactions: warmth, discomfort, acne (Skin and subcutaneous tissue disorders) | 11 (14)
Headache/ Migraines (General disorders) | 9 (12)
Flu/cold like symptoms: sore throat, sinusitis, post nasal drip (Infections and infestations) | 12 (13)
Sleep-related: insomnia, early insomnia, nightmare, sleep talking, vivid dreams (General disorders) | 9 (10)
Gastrointestinal: acute GE, heartburn (Gastrointestinal disorders) | 2 (2)
Mood symptoms: anhedonia, depressed symptoms, school anxiety, separation anxiety (Psychiatric disorders) | 4 (4)
Other: fatigue, redness on cheeks, sweating, eye pain, toothache, nosebleed (General disorders) | 7 (8)
Allergies, Itch (Immune system disorders) | 2 (2)
Iritability/ distractibility (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/58/NCT04569058/Prot_SAP_000.pdf